CLINICAL TRIAL: NCT03240107
Title: Standard Levator Aponeurosis / Muscle Resection With Three Point Fixation Versus Two Point Fixation Tucking for Congenital Ptosis With Fair to Good Levator Function
Brief Title: Levator Resection with3 Point Fixation Versus 2 Point Fixation Tucking for Congenital Ptosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heba Hamdy Ibrahim Mohammed (Other)
Responsible Party: Sponsor-Investigator, Heba Hamdy Ibrahim Mohammed, Doctor heba hamdy ibrahim, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hhim123
Record Dates: First submitted 2016-12-16; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-07

CONDITIONS: Congenital Ptosis
Keywords: levator resection; levator tucking; Fair levator function; Eyelid contour

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levator resection (Active Comparator): 20 patients who will undergo levator aponeurosis resection technique
  Interventions: Procedure: levator resection
- levator tucking (Active Comparator): 20 patients who will undergo two point fixation levator tucking technique
  Interventions: Procedure: levator tucking

INTERVENTIONS:
Procedure: levator resection — The levator aponeurosis was dissected from the upper border of the tarsal plate and conjunctiva.
  The aponeurosis was measured for the desired amount of resection and fixed to the exposed tarsal border with three point mattress sutures with 6-0 prolene then amount measured resect.
  The skin incision closed by continuous suture with 6-0 prolene.
  Arms: levator resection
Procedure: levator tucking — The levator aponeurosis was dissected from the upper border of the tarsal plate and conjunctiva.
  . The aponeurosis was measured for desired amount of tucking The skin incision closed by continuous suture with 7-0 prolene.
  Arms: levator tucking

SUMMARY:
to evaluate the surgical effect of levator aponeurosis resection Versus two point fixation levator aponeurosis Tucking for Congenital Ptosis

DETAILED DESCRIPTION:
Target population for the study is children under twelve years old presenting to ophthalmology clinic at Cairo university specialized pediatric hospital with congenital ptosis.

Patients will be randomly divided into two groups First group (A) will contain 20 patients who will undergo standard levator aponeurosis resection Second group (B) will contain 20 patient who will undergo two point fixation levator tucking

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral or bilateral simple isolated congenital ptosis.
2. Levator function more than 4mm

Exclusion Criteria:

1. Congenital ptosis associated with other ocular syndromes.
2. Recurrent ptosis following any attempt for repair.
3. Traumatic ptosis or acquired ptosis
4. -ve bell's phenomenon.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Comparison of surgical efficacy of standard levator aponeurosis resection and two point fixation tucking regarding MRD1 | 6 to 9 months
  MRD1:distance between upper lid margin and corneal light reflex measured in mm by transparent ruler

CONTACTS AND LOCATIONS:
Overall Officials: RANIA AS EL ASSAWY, PhD, Study Chair — Cairo University; Sameh HA ABDEL BAKY, MD, Study Director — Cairo University; DINA HO HASSANIEN, MD, Study Director — Cairo University
Locations (1):
- HEBA, Cairo, Zahraa AL Maadi, Egypt

IPD SHARING:
Plan to Share IPD: Undecided